CLINICAL TRIAL: NCT05888493
Title: A Randomized, Open-label, Multi-center Phase III Trial Comparing Tisagenlecleucel to Standard of Care in Adult Participants With Relapsed or Refractory Follicular Lymphoma (FL)
Brief Title: A Phase III Trial Comparing Tisagenlecleucel to Standard of Care (SoC) in Adult Participants With r/r Follicular Lymphoma
Acronym: LEDA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCTL019E2301; 2023-503452-27-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-05-01; First posted 2023-06-05 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Follicular Lymphoma (FL)
Keywords: relapsed or refractory follicular lymphoma; r/r; FL; CAR-T; tisagenlecleucel; CTL019; phase III; standard of care; SOC
MeSH Terms: conditions — Lymphoma, Follicular; Recurrence | interventions — tisagenlecleucel; Lenalidomide; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Prednisolone; R-CHOP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tisagenlecleucel (Experimental): Participants randomized to the tisagenlecleucel treatment strategy will receive a single infusion of 0.6 to 6 x 10^8 CAR-positive viable T-cells
  Interventions: Biological: Tisagenlecleucel; Drug: Lymphodepleting chemotherapy; Other: Corticosteroids and/or Radiation (Bridging therapy)
- R2 or R-CHOP (Active Comparator): Participants randomized to Standard of Care treatment will receive either R2 or R-CHOP based on investigator choice of therapies, and this has to be determined prior to randomization.
  Interventions: Drug: Lenalidomide and rituximab (R2) in 28-day cycles for up to 12 cycles.; Drug: Rituximab, cyclophosphamide, doxorubicin, vincristine and prednisone or prednisolone (R-CHOP) in 21-day cycles for 6 to 8 cycles

INTERVENTIONS:
Biological: Tisagenlecleucel — Tisagenlecleucel is a solution for infusion of 0.6 to 6 x 10^8 CAR-positive viable T-cells taken intravenously (i.v.).
  Other Names: CTL019
  Arms: Tisagenlecleucel
Drug: Lenalidomide and rituximab (R2) in 28-day cycles for up to 12 cycles. — Lenalidomide 20 mg daily on days 1-21 for up to 12 cycles Rituximab 375 mg/m2 IV on days 1, 8, 15, and 22 of cycle 1 and day 1 of cycles 2-5
  Other Names: R2
  Arms: R2 or R-CHOP
Drug: Rituximab, cyclophosphamide, doxorubicin, vincristine and prednisone or prednisolone (R-CHOP) in 21-day cycles for 6 to 8 cycles — Rituximab 375 mg/m2 i.v. on day 1 Cyclophosphamide 750 mg/m2 i.v. day 1 Doxorubicin 50 mg/m2 i.v. day 1 Vincristine 1.4 mg/2 (capped at 2 mg) i.v. day 1 Prednisone or prednisolone 40 mg/m2 PO days 1-5
  Other Names: R-CHOP
  Arms: R2 or R-CHOP
Drug: Lymphodepleting chemotherapy — Fludarabine (25 mg/m^2 intravenously [i.v.] daily for 3 doses) OR Cyclophosphamide (250 mg/m^2 i.v. daily for 3 doses starting with the first dose of fludarabine).
  OR Bendamustine 90 mg/m^2 i.v. daily for 2 days (If there was previous grade IV hemorrhagic cystitis with cyclophosphamide, or the participant demonstrated resistance to a previous cyclophosphamide-containing regimen)
  Arms: Tisagenlecleucel
Other: Corticosteroids and/or Radiation (Bridging therapy) — Corticosteroids and/or Radiation
  Arms: Tisagenlecleucel

SUMMARY:
This trial will compare tisagenlecleucel to standard of care in adult participants with relapsed or refractory (r/r) follicular lymphoma.

DETAILED DESCRIPTION:
The purpose of this phase III study is to verify the clinical benefit of tisagenlecleucel for the treatment of r/r FL by comparing the tisagenlecleucel treatment strategy to standard of care therapy in patients with r/r FL after two or more lines of systemic therapy, with progression-free survival (PFS) as the primary endpoint.

The primary objective is to demonstrate superiority of the tisagenlecleucel treatment strategy over standard of care (SOC) therapy with respect to progression-free survival (PFS) determined by blinded independent review committee (BIRC) based on the Lugano response criteria.

Participants randomized to Arm A (tisagenlecleucel treatment) will receive a single infusion of 0.6 to 6 x 10^8 CAR-positive viable T-cells.

Participants randomized to Arm B (Standard of Care) will receive R2 or R-CHOP based on investigator choice and this has to be determined prior to randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the date of signing the informed consent form.
2. Follicular lymphoma grade 1, 2, or 3A confirmed histologically after latest relapse (local assessment).
3. Relapsed or refractory disease after a second or later line of systemic therapy including an anti-CD20 antibody and an alkylating agent.
4. Disease that is both active on Positron emission tomography (PET) scan (defined as a score of 4 or 5 on the Deauville 5-point scale) and measurable on Computed tomography (CT) scan.
5. ECOG performance status of 0, 1 or 2 at screening.
6. Adequate hematologic, renal, hepatic and pulmonary organ function at screening.
7. Must meet the institutional criteria to undergo leukapheresis (unless historical leukapheresis is available).
8. Must be eligible for treatment with the selected standard of care regimen.

Exclusion Criteria:

1. Follicular lymphoma grade 3B or evidence of histologic transformation.
2. Prior treatment with anti-CD19 therapy, gene therapy, or adoptive T-cell therapy.
3. Active CNS involvement by malignancy.
4. Clinically significant active infection, presence of Human immunodeficiency virus (HIV) antibody or active hepatitis B or C.
5. Active neurological autoimmune or inflammatory disorders (e.g., Guillain-Barré syndrome).
6. Investigational medicinal product within the last 30 days or five half-lives (whichever is longer) prior to randomization.
7. Clinically significant cardiovascular conditions such as acute coronary syndrome, significant cardiac arrhythmias, heart failure or decreased LVEF.

Other protocol defined inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2028-07-25 (Estimated); Study Completion 2031-01-18 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) determined by blinded independent review committee (BIRC) | 5 years
  Progression free survival (PFS) based on Lugano response criteria, defined as time from randomization to the first of the following events to occur:
  * progressive disease (by BIRC)
  * death from any cause

SECONDARY OUTCOMES:
Complete response rate (CRR) as assessed by BIRC (Key Secondary) | 5 years
  CRR: The proportion of participants with BOR of complete response (CR)
Overall response rate (ORR) by BIRC | 5 years
  ORR: The proportion of participants with BOR of either CR or partial response (PR)
Overall survival (OS) | 5 years
  OS: Time from randomization to date of death due to any cause
Time to next anti-lymphoma treatment (TTNT) | 5 years
  TTNT: Time from randomization until start of new anticancer therapy or death due to any cause.
Duration of Response (DOR) | 5 years
  Time from the date of first documented BIRC response of CR or PR to the date of first documented progression by BIRC or any cause of death
Pre-existing (prior to treatment) and treatment-induced anti-mCAR antibodies (humoral immunogenicity) | 5 years
  Summarize percentage of patients with pre-existing and treatment-induced anti-mCAR antibodies, and relate the antibody responses with CAR expansion, efficacy, and safety endpoints.
CAR transgene levels, as measured by quantitative polymerase chain reaction (qPCR), in peripheral blood, bone marrow (and other tissues, if available) | 5 years
  Summary of transgene levels by timepoints and by clinical responses, cellular kinetic parameters will be derived using non-compartmental analysis from time course of transgene levels and will be summarized by clinical responses.
Replication competent lentivirus (RCL) by VSV-g qPCR in participants receiving tisagenlecleucel | 5 years
  This is to assess presence of (Replication competent lentivirus) RCL in participants receiving tisagenlecleucel by VSV-g qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (32):
- United States (2):
  - TRIHEALTH Good Samarithan Hospital, Cincinnati, Ohio
  - VA Tennessee Valley Healthcare System, Nashville, Tennessee
- Australia (4):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Austria (2):
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Ostrava, Poruba, Czechia
- Novartis Investigative Site, Budapest, Hungary
- Poland (4):
  - Novartis Investigative Site, Poznan, Greater Poland Voivodeship
  - Novartis Investigative Site, Gliwice, Silesian Voivodeship
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Lodz
- Novartis Investigative Site, Bucharest, Romania
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Bratislava, Slovakia
- Novartis Investigative Site, Seoul, South Korea
- Spain (9):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Madrid
- Taiwan (3):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com